CLINICAL TRIAL: NCT04998461
Title: Impact of Obesity, Chronic Kidney Disease and Type 2 Diabetes on Human Urinary Stem Cells
Acronym: URISTEM
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0907; 2021-A02135-36 (Other: ID-RCB)
Record Dates: First submitted 2021-08-02; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Chronic Kidney Diseases; Obesity; Stem Cells; Diabetes type2
Keywords: bio-marker; Chronic Kidney Diseases; Obesity; Diabetes type2
MeSH Terms: conditions — Renal Insufficiency, Chronic; Obesity | interventions — Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Obese patients with normal renal function: * estimated Glomerular Filtration Rate (eDFG) ≥ 60 ml/min/1.73 m2
  * Body Mass Index (BMI) > 30 kg/m2
  * Microalbuminuria / creatinuria ≤ 3mg / mmol and / or proteinuria < 0.15 g/24h
  Interventions: Biological: urine collection
- Obese patients with impaired renal function: * estimated Glomerular Filtration Rate (eDFG) < 60 ml/min/1.73 m2
  * Body Mass Index (BMI) > 30 kg/m2
  * Microalbuminuria / creatinuria ≤ 3mg / mmol and / or proteinuria < 0.15 g/24h
  Interventions: Biological: urine collection
- Non-obese patients with impaired renal function: * estimated Glomerular Filtration Rate (eDFG) < 60 ml/min/1.73 m2
  * Body Mass Index (BMI) between 18 and 30 kg/m2
  * Microalbuminuria / creatinuria ≤ 3mg / mmol and / or proteinuria < 0.15 g/24h
  Interventions: Biological: urine collection
- Non-obese patients with normal renal function (control group): * estimated Glomerular Filtration Rate (eDFG) ≥ 60 ml/min/1.73 m2
  * Body Mass Index (BMI) between 18 and 30 kg/m2
  * Microalbuminuria / creatinuria ≤ 3mg / mmol and / or proteinuria < 0.15 g/24h
  Interventions: Biological: urine collection

INTERVENTIONS:
Biological: urine collection — To isolate urine stem cells, a sample of 30ml minimum an 100ml maximum as a function of the patient, will be collected in a single time in a sterile flask during collection for the nephrologic exams. A transcriptome analysis of USC will be performed.

SUMMARY:
Obesity is at risk for the development of chronic kidney disease but the involved mechanisms are not known (Navarro et al. 2015). Establishing the link between obesity and kidney damage is difficult. Indeed, kidney function measurement lacks precision in obese people (Lemoine et al. 2014) and requires expensive methods such as measurement of 99mTc-DTPA clearance. Biopsies are too invasive for the detection of emerging kidney damage or for the following of the kidney function. Therefore new tools are required for the early identification of at risk individuals for the kidney damage complication.

Mesenchymal stem cells may represent such a relevant tool. These cells are present in a large number of organs, including kidney (Costa et al. 2020).

In addition to be differentiated cells progenitors (Dominici et al. 2006), they also support immunosuppressive, anti-fibrotic and pro-angiogenic functions that have been used for the treatment of kidney fibrosis (Usunier et al. 2014). Therefore, mesenchymal stem cells contribute to tissue homeostasis and their alterations may reflect organ dysfunctions. Indeed, mesenchymal stem cells from obese adipose tissue lose their immunosuppressive (Serena et al. 2016) and differentiation (Gustafson et al. 2009) functions and contribute to fibrosis (Keophiphath et al. 2009) and inflammation (Lee et al. 2010; Gustafson, Nerstedt, et Smith 2019). It is thus probable that kidney dysfunctions are associated with functional alterations of kidney mesenchymal stem cells.

The collection of mesenchymal stem cells from kidney can easily be performed from urine and next cultivated for amplification. They are called urine stem cells (USC).

From our experience with obese mouse adipose stem cells, we observed that functional changes of stem cells preceded adipose tissue dysfunctions. Functional signatures of mesenchymal stem cells are thus representative of changes occuring in the function of the tissue notably in answer to obesity. These features could be used to identify obese people presenting ongoing alterations of kidney function, before clinical manifestations of kidney dysfunction. Because kidney mesenchymal stem cells are easy to isolate from urine, their collection is compatible with the follow up of patients and can be applied to a large number of individuals, including the younger. USC could represent a valuable tool to detect progression towards kidney damage.

In this project we plan to analyse USC alterations induced by obesity and to identify signatures associated with the progression towards kidney damage and type 2 diabetes. The goal is to evaluate USC as potential marker for the non invasive monitoring of patients in answer to a need that is not achieved by the present available approaches.

ELIGIBILITY:
Inclusion Criteria - For all participants :

* Age between 18 and 60
* Non diabetic (fasting blood glucose <1.26 g/L)
* Patient not having objected to participating in the research

Inclusion Criteria - For the obese group with normal renal function

* eDFG ≥ 60 ml/min/1.73 m2
* BMI > 30 kg/m2
* Microalbuminuria / creatinuria ≤ 3mg / mmol and / or proteinuria < 0.15 g/24h

Inclusion Criteria - For the obese group with impaired renal function

* eDFG < 60 ml/min/1.73 m2
* BMI > 30 kg/m2
* Microalbuminuria / creatinuria ≤ 3mg / mmol and / or proteinuria < 0.15 g/24h

Inclusion Criteria - For the non-obese group with impaired renal function

* eDFG < 60 ml/min/1.73 m2
* BMI between 18 and 30 kg/m2
* Microalbuminuria / creatinuria ≤ 3mg / mmol and / or proteinuria < 0.15 g/24h

Inclusion Criteria - For the non-obese group with normal renal function (control group)

* eDFG ≥ 60 ml/min/1.73 m2
* BMI between 18 and 30 kg/m2
* Microalbuminuria / creatinuria ≤ 3mg / mmol and / or proteinuria < 0.15 g/24h

Exclusion Criteria - For all participants :

* Acute renal failure within 3 months (defined as an increase of more than 50% in usual creatinemia)
* Inflammatory, infectious, cardiovascular or progressive neoplastic disease
* Urinary pathology (malformation, infection, etc.)
* Exclusion period of a previous study or already participating in a clinical research protocol having an impact on the judgment criteria of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will focus on 4 groups of non-diabetic patients, namely:
  1. obese patients with preserved renal function
  2. obese patients with renal failure
  3. non-obese patients with preserved renal function
  4. non-obese patients with renal failure (study control group)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of gene expression in USC (Urinary Stem Cells) | inclusion day
  High throughput sequencing will be used to compare USC (Urinary Stem Cells) for the differential expression of genes between the 4 populations (obese or lean patients, with or without alteration of the kidney function). A gene set enrichment analysis will be used to identify the main functions supported by USC from each patient, establishing a signature.

CONTACTS AND LOCATIONS:
Overall Officials: Laetitia KOPPE, PhD, Principal Investigator — Service de néphrologie
Locations (1):
- Centre Hospitalier Lyon SUD, Pierre-Bénite, France